CLINICAL TRIAL: NCT04326673
Title: Salivary Testosterone in Men: Diurnal Variation and Post-prandial Responses
Acronym: SalT
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020LAB110
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Hypogonadism, Male
MeSH Terms: conditions — Eunuchism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diurnal variation assessment: Assessment of diurnal variation in salivary testosterone adjusted for prandial state
  Interventions: Other: Testosterone Measurements in healthy volunteers after fasting
- Glucose load measurements: Measurement of salivary and serum testosterone and related biomarkers before and after a standard 75g oral glucose load
  Interventions: Other: Testosterone Measurements after glucose loading

INTERVENTIONS:
Other: Testosterone Measurements in healthy volunteers after fasting — salivary testosterone measurements taken in morning and evening and a single blood test for testosterone taken
  Groups: diurnal variation assessment
Other: Testosterone Measurements after glucose loading — salivary tstosterone and blood testosterone measurements
  Groups: Glucose load measurements

SUMMARY:
The purpose is to evaluate Sal-T against standard biomarkers of male gonadal status based on serum T, calculated free T and BAT. The optimal salivary sampling in terms of fasting and time of day will also be defined.

The ultimate aim is to add Sal-T into the Trust's repertoire of tests in investigating suspected hypogonadism in men.

DETAILED DESCRIPTION:
To investigate whether salivary (free) testosterone is subject to similar prandial variations reported for serum total testosterone.

Study 1:

Assessment of diurnal variation in salivary testosterone adjusted for prandial state in 20 healthy men.

Study 2:

Measurement of salivary and serum testosterone and related biomarkers before and after a standard 75g oral glucose load in 40 men.

ELIGIBILITY:
For 1st part of study -volunteers:

Inclusion Criteria:

* Aged 20-60 years
* Male

Exclusion Criteria:

* Subjects with learning disability or those lacking mental capacity to give consent.
* On (prescribed and over-the-counter) medication and herbal remedies known to affect androgen metabolism.
* Known hypogonadism.
* Conditions known to affect androgen metabolism, including chronic inflammatory diseases, chronic liver disease, chronic kidney disease and thyroid dysfunction.
* Any co-morbidity.
* Periodontal disease.
* Dental work 48 hours prior to the test.
* Exercise on the day, prior to and during sampling periods.
* Brushed teeth within 1hr prior to sample collection.
* Obesity defined as a body mass index (BMI) of greater than 29.9 kg/m2As

  2nd part of study for glucose load - oral glucose tolerance test (OGTT):

Inclusion criteria:

* Aged over 40-60 years.
* Attending for routine 75 g OGTT

Exclusion criteria:

* Subjects with learning disability or lacking mental capacity to give consent.
* On (prescribed and over-the-counter) medication and herbal remedies known to affect androgen metabolism.
* Known hypogonadism.
* Conditions known to affect androgen metabolism, including chronic inflammatory diseases, chronic liver disease, chronic kidney disease and thyroid dysfunction.
* Subjects with difficult venous access.
* Periodontal disease.
* Dental work 48 hours prior to the test.
* Brushed teeth within 1hour prior to sample collection.
* Exercise on day prior to and during the OGTT.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers and patients attending hospital for their OGTT as part of their stnadard care.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Changes in salivary testosterone during the day independent of prandial state | 24 hours
  testosterone levels
Changes in salivary testosterone following an oral glucose load | 2 hours
  testosterone levels

CONTACTS AND LOCATIONS:
Overall Officials: R Gama, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fenn J, Gill H, Starbrook L, Ford L, Sharrod-Cole H, Kalaria T, Ford C, Gama R. Salivary testosterone changes during oral glucose tolerance tests in overweight and obese men - Postprandial or circadian variation? Ann Clin Biochem. 2024 Sep;61(5):391-398. doi: 10.1177/00045632241249087. Epub 2024 May 9. PMID 38591370